CLINICAL TRIAL: NCT01309178
Title: Anti-inflammatory Pulmonal Therapy of CF Patients With Amitriptyline and Placebo - a Randomised, Double-blind, Placebo-controlled, Multicenter, Cohort - Study
Brief Title: Anti-inflammatory Pulmonal Therapy of Cystic Fibrosis (CF) Patients With Amitriptyline and Placebo
Acronym: APA-IIb
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Children's Hospital Tuebingen (Other)
Collaborators: Universität Duisburg-Essen (Other); University of Ulm (Other)
Responsible Party: University Hospital Tuebingen, University Children´s Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APA-IIb; 2008-002673-13 (EudraCT Number)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2009-03

CONDITIONS: Cystic Fibrosis; Pneumonia
MeSH Terms: conditions — Cystic Fibrosis; Pneumonia | interventions — Amitriptyline; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amitriptyline (Active Comparator): After the experience with the treatment of 18 CF-patients phase IIa study), the medication will be therefore 25 mg daily in two doses (2 x 12,5 mg). Because of a higher rate of side effects (tiredness, dry mucous membrane) the higher dose of 50 mg (2 x 25 mg) is not chosen first, but will be adapted after 2 weeks of treatment.
  Interventions: Drug: Amitriptyline
- Mannite (Placebo Comparator): The placebo will be given 25 mg daily in two doses (2 x 12,5 mg). After 2 weeks of treatment the higher dose of 50 mg (2 x 25 mg) will be given
  Interventions: Drug: Mannite

INTERVENTIONS:
Drug: Amitriptyline — 2 x 12,5 mg capsules for oral use in the first two weeks, the higher dose of 50 mg (2 x 25 mg) will be adapted after 2 weeks of treatment.
  Other Names: Amitriptylinhydrochlorid
  Arms: Amitriptyline
Drug: Mannite — Mannit capsules daily in two doses (2 x 12,5 mg). After 2 weeks of treatment the higher dose of 50 mg (2 x 25 mg) will be given
  Other Names: Mannite Ph. Eur.
  Arms: Mannite

SUMMARY:
Cystic fibrosis patients suffer from a chronic destruction of the lung, frequent and finally chronic pneumonia and a reduced life expectancy. Unfortunately, no curative treatment for cystic fibrosis is available, neither are treatments established that prevent the disease. Our data identify ceramide as a potential novel target to treat cystic fibrosis.

Two smaller trials support the notion that inhibition of the acid sphingomyelinase by amitriptyline improves the lung function of CF-patients even at a dose that is low enough to avoid adverse effects.

In the present proposal the investigators, therefore, aim to test in a larger cystic fibrosis patient population whether an inhibition of ceramide release in the lung caused by the lack of functional CFTR improves the lung function of cystic fibrosis patients. Inhibition of ceramide-release in the lung will be achieved by treatment with amitriptyline, which is used as an anti-depressant drug for almost 50 years. Although it is not absolutely specific, it seems to be relatively specific for the degradation of acid sphingomyelinase (typically 60-80% of cellular acid sphingomyelinase are degraded), which releases ceramide from sphingomyelin.

If the data confirm the beneficial effect of amitriptyline already observed in our preliminary studies, the present clinical study may establish a novel treatment to improve clinical symptoms of cystic fibrosis and, moreover, to prevent or at least delay the onset of cystic fibrosis.

Hypothesis

* Amitriptyline reduces ceramide concentrations in respiratory epithelial cells (measured in nasal epithelial cells obtained by brushing nasal mucosa).
* Amitriptyline treatment reduces cell death in bronchi and deposition of DNA on the respiratory epithelium, which permits elimination of P. aeruginosa from the lung (measured as P. aeruginosa counts in tracheal fluid).
* Amitriptyline treatment results in normalization of the function of leukocytes (number determined in serum and tracheal fluid)
* Amitriptyline reduces systemic and local inflammation (measured as cytokines in plasma and tracheal fluid).

Based on these effects amitriptyline increases the lung function of cystic fibrosis patients (measured by FEV1).

DETAILED DESCRIPTION:
Cystic fibrosis (CF), the most common autosomal recessive disorder at least in western countries, is caused by mutations of the cystic fibrosis transmembranous conductance regulator molecule (CFTR) and affects approximately 40 000 patients in Europe. Most, if not all, CF-patients develop a chronic pulmonary infection with Pseudomonas aeruginosa (P. aeruginosa). At present, it is unknown why CF-patients are highly sensitive to P. aeruginosa infections and, most importantly, no curative treatment for cystic fibrosis is available.

Our studies provided a novel pathophysiological concept for cystic fibrosis. The investigators demonstrated that ceramide plays a crucial role in the development of cystic fibrosis and the high sensitivity of Cftr-deficient mice to infection with P. aeruginosa (1,2). Using biochemical techniques, fluorescence microscopy, and mass spectrometry, the investigators found that ceramide accumulates in the lungs of various Cftr-deficient mouse strains before any infection occurs, in particular in the epithelial cells of large and small bronchi and in alveolar macrophages. The accumulation of ceramide in Cftr-deficient epithelial cells may be mediated by an increase in pH from 4.5 to 6.0 in secretory lysosomes and pre-lysosomes of Cftr-deficient cells. The change in pH results in a reduction of approximately 90% in the activity of acid ceramidase which consumes ceramide, and a reduction of only 35% in the activity of acid sphingomyelinase which releases ceramide. An imbalance in the activity of these two enzymes, by which a relative over-activity of acid sphingomyelinase produces ceramide, may then result in an accumulation of ceramide. Partial inhibition of acid sphingomyelinase, either genetically or pharmacologically, returns ceramide concentrations to near normal levels in the lungs of Cftr-deficient mice. Genetic inhibition of acid sphingomyelinase was achieved by crossing Cftr-deficient mice with acid sphingomyelinase-deficient mice to create mice deficient in Cftr and heterozygous for acid sphingomyelinase (Cftr-/-/Smpd1+/- mice). The activity of acid sphingomyelinase in the lungs of these mice was approximately 50% lower than in the lungs of wild-type mice. Pharmacological inhibition of acid sphingomyelinase was achieved by treating Cftr-deficient mice with the functional acid sphingomyelinase inhibitor amitriptyline (1,2). Increased concentrations of ceramide in the bronchial epithelial cells of Cftr-deficient mice triggered death of these cells, the deposition of DNA in bronchi, chronic pulmonary inflammation, and a high susceptibility of Cftr-deficient mice to pulmonary infections with P. aeruginosa. Normalisation of ceramide concentrations by genetic means normalised these changes, and pharmacological inhibition of acid sphingomyelinase prevented these changes. Ceramide accumulation was also observed in ciliated nasal epithelial cells, macrophages and lung transplant materials from CF patients (1-4). This finding suggests that the results of our murine studies also apply to humans with cystic fibrosis. Next, the investigators applied a panel of functional inhibitors of acid sphingomyelinase and treated Cftr-deficient mice by inhalation of amitriptyline, trimipramine, desipramine, chlorprothixene, fluoxetine, amlodipine, or sertraline, all of which are functional inhibitors of acid sphingomyelinase. This inhalation reduced the activity of acid sphingomyelinase specifically in the lung and normalised pulmonary ceramide concentrations, inflammation, and susceptibility to infection (2). Recent findings by C. Ward and associates confirmed the accumulation of ceramide in lung specimens from CF patients (5).

Clinical data:

1. Pilot study - Based on the amitriptyline-mediated protection of Cftr-deficient mice, the investigators initiated a small clinical cross over study with 4 cystic fibrosis patients that were treated with amitriptyline or placebo, respectively. The results revealed a clinical relevant increase of the lung function (determined as FEV1) in all cystic fibrosis patients after treatment with amitriptyline for 2 weeks.
2. Phase IIa - The positive data of the pilot study encouraged us to initiate a Phase IIa cross over study in 18 patients and to investigate a beneficial effect of amitriptyline on cystic fibrosis in a larger patient population to prove safety, biochemically prove the mechanisms of action, and for dose finding of amitriptyline (25 mg/day, 50 mg/day, 75 mg/day). Amitriptyline was well-tolerated in the patient group and no SAEs were recorded at the end of the 28-day-course. From the 80 AEs, 35 were related or possibly related to the medication. Two well-known AEs of amitriptyline, i.e. xerostomia and tiredness, were significantly different between placebo and the three amitriptyline treatment groups, but were mostly transient. FEV1 was analysed in the per protocol analysis in 13, 7, 8 and 8 available patient cycles, who had received placebo, 25 mg, 50 mg or 75 mg amitriptyline/day, respectively. After 14 days of treatment the primary endpoint FEV1 had improved significantly in the 25 mg/d amitriptyline group relative to placebo (FEV1: +5.0% compared to the placebo group; p = 0.048). No significant change of lung function was observed when patients were administered 50 mg and 75 mg of amitriptyline (6).
3. Phase IIb - To evaluate the positive data of the phase IIa-trial, the investigators initiated a phase IIb study in 2009 with a parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis is verified
* Patient is older than 14 years
* Patients weight is more than 35 kg
* FEV1 is higher than 30% and lower than 90%
* The patient is pulmonal colonized with bacteria
* No acute pulmonal illness is present
* CRP is not elevated two fold (2 mg/dl) of normal
* Lung function testing is possible
* A full course of therapy is possible without any restrictions

Exclusion Criteria:

* FEV1 in baseline differs more than 10% from screening visit
* CRP in baseline differs more than 50% from screening visit
* Glaucoma, seizures, heart insufficiency or major depression are present
* Intravenous antibiotic treatment was necessary in the last 4 weeks before visit 2
* High dose steroid therapy
* On-off-therapy of tobramycin in the last 2 weeks
* Involvement of the patient in another study
* Pregnancy and
* Nursing mothers

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of the lung function parameter FEV1 (absolute and relative to baseline) under verum and placebo | in 4 weeks
  The primary aim is the change of the lung function parameter Forced Expiratory Volume in 1 second (FEV1) relative to baseline under verum and placebo

SECONDARY OUTCOMES:
Increase in lung function measurements | in 2 and 4 weeks
  Increase (absolute and relative to baseline) in lung function (FVC, FEV1, MEF 25, LCI, CO-Diffusion) in 2 and 4 weeks
Ceramide concentration in epithelial cells | in 4 weeks
  Decrease of Ceramide concentration in epithelial cells detected in sputum
Inflammation status | in 4 weeks
  Reduction of IL-8 (facultatively IL-1ß, IL-6, IL-8, TNFα) as well as an increase of anti-inflammatory IL-10 in tracheal mucus
Bacteriological and cell status | in 4 weeks
  Reduction of the DNA-content and granulocyte concentration and decrease of chronic bacterial colonization (P. aerug., S. aureus, etc.) in tracheal mucus.
Side effects | in 4 weeks
  Number of upper and lower respiratory tract infections pulmonary exacerbations)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Riethmueller, Dr, Study Director — University Children´s Hospital Tubeingen, Germany
Locations (3):
- Germany (3):
  - Lutz Naehrlich, Giessen
  - Jochen Mainz, Jena
  - Joachim Riethmueller, Tübingen